CLINICAL TRIAL: NCT05747027
Title: Prospective Randomized Controlled Trial Comparing Transvaginal Rectopexy and Ventral Mesh Rectopexy for Obstructed Defecation in Pelvic Organ Prolapse (PROD Trial)
Brief Title: Prospective Randomized Controlled Trial of Obstructed Defecation Surgery
Acronym: PROD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low recruitment rate
Sponsor: Endeavor Health (Other)
Collaborators: Weill Medical College of Cornell University (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Ghazaleh Rostami Nia, Director of Research Division of Urogynecology, NorthShore University HealthSystem, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EH22-284
Record Dates: First submitted 2023-02-05; First posted 2023-02-28 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Obstructed Defecation; Pelvic Organ Prolapse
Keywords: Rectopexy; Transvaginal rectopexy; Laparoscopic ventral rectopexy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Masking Description: The study surgeon is providing clinical care to enrolled subjects, thus masking the surgeon to treatment allocation or subject symptoms is not practical or feasible, other than the allocation concealment prior to surgical randomization. Given the surgical procedure requires a transvaginal or abdominal incision, it is clinically not possible to mask the participant or other research personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic abdominal ventral rectopexy (Experimental)
  Interventions: Procedure: Laparoscopic abdominal ventral rectopexy
- Transvaginal sacrospinous rectopexy (Experimental)
  Interventions: Procedure: Transvaginal sacrospinous rectopexy

INTERVENTIONS:
Procedure: Laparoscopic abdominal ventral rectopexy — Laparoscopic abdominal ventral rectopexy is an established surgical technique used to restore rectal support in women with obstructive defecatory syndrome (ODS). It is the most common surgery used to treat ODS. It involves a series of small cuts in the abdomen and the use of mesh to hold the rectum in the correct position.
  Arms: Laparoscopic abdominal ventral rectopexy
Procedure: Transvaginal sacrospinous rectopexy — Transvaginal sacrospinous rectopexy is an innovative procedure which has shown to be safe and effective in the treatment of stool entrapment. This is a mesh-free and vaginal route procedure.
  Arms: Transvaginal sacrospinous rectopexy

SUMMARY:
Obstructive defecatory syndrome (ODS) or inability to completely empty bowel is characterized by a combination of straining, incomplete evacuation, and the use of digital manipulation with bowel movement. This is a common condition with estimated incidence of 15-20% in the adult female population.

Laparoscopic abdominal ventral rectopexy is an established surgical technique aimed at restoring rectal support in women with this condition. It is the most common surgery used nowadays to treat ODS. Transvaginal sacrospinous rectopexy, is an innovative procedure which has been shown to be safe and effective in the treatment of stool entrapment. Currently it is unknown whether one of the procedures mentioned is superior to the other regarding surgical outcomes and patient experience. The purpose of this research is to compare the outcomes of these two procedures considering their efficacy to improve symptoms.

During the study, participants will be randomized to undergo one of two procedures for treatment of inability to completely empty their bowel and/or rectal prolapse: 1) laparoscopic abdominal ventral rectopexy; 2) transvaginal sacrospinous rectopexy. Following the procedure, participants will be asked to return to the office for a follow-up visit 2-weeks, 2-, 12- and 24-months after the surgery. During each follow-up visit participants will undergo symptom evaluation, pelvic exam and transvaginal pelvic ultrasound to evaluate surgical success.

ELIGIBILITY:
Inclusion Criteria:

1. Female, between the age of 18 and 80
2. OD symptoms as indicated by an affirmative response to either questions 7, 8 or 14 of the Pelvic Floor Distress Inventory (PFDI):

   1. Do you feel you need to strain too hard to have a bowel movement?
   2. Do you feel you have not completely emptied your bowels at the end of a bowel movement?
   3. Does part of your bowel ever pass through the rectum and bulge outside during or after a bowel movement?
3. Rectal hypermobility defined as a compression ratio greater than 50% according to ultrasound
4. Patient planning on undergoing surgery for the repair of pelvic organ prolapse within the next 12 months
5. Patient who is not pregnant and does not intend to become pregnant in the next 2 years
6. Available for 24-months of follow-up
7. Stated willingness to comply with all study procedures and availability for the duration of the study
8. Able to complete study assessments, per clinician judgment
9. Able and willing to provide independent written informed consent
10. Stable cardiovascular and respiratory status to meet candidacy in vaginal or laparoscopic surgeries

Exclusion Criteria:

1. Contraindication to abdominal and transvaginal rectopexy in the opinion of the treating surgeon
2. History of previous surgery that included any type of surgery for rectal prolapse
3. Pelvic pain or dyspareunia due to levator ani spasm that would preclude a PMT program
4. Previous adverse reaction to synthetic mesh
5. Current cytotoxic chemotherapy or current or history of pelvic radiation therapy within 12 months
6. History of two inpatient hospitalizations for medical comorbidities in the previous 12 months

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ghazaleh Rostami Nia, MD, Principal Investigator — Endeavor Health
Locations (2):
- United States (2):
  - Endeavor Health, Skokie, Illinois
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bove A, Pucciani F, Bellini M, Battaglia E, Bocchini R, Altomare DF, Dodi G, Sciaudone G, Falletto E, Piloni V, Gambaccini D, Bove V. Consensus statement AIGO/SICCR: diagnosis and treatment of chronic constipation and obstructed defecation (part I: diagnosis). World J Gastroenterol. 2012 Apr 14;18(14):1555-64. doi: 10.3748/wjg.v18.i14.1555. PMID 22529683
- [Background] Bove A, Bellini M, Battaglia E, Bocchini R, Gambaccini D, Bove V, Pucciani F, Altomare DF, Dodi G, Sciaudone G, Falletto E, Piloni V. Consensus statement AIGO/SICCR diagnosis and treatment of chronic constipation and obstructed defecation (part II: treatment). World J Gastroenterol. 2012 Sep 28;18(36):4994-5013. doi: 10.3748/wjg.v18.i36.4994. PMID 23049207
- [Background] Lembo A, Camilleri M. Chronic constipation. N Engl J Med. 2003 Oct 2;349(14):1360-8. doi: 10.1056/NEJMra020995. No abstract available. PMID 14523145
- [Background] D'Hoore A, Penninckx F. Obstructed defecation. Colorectal Dis. 2003 Jul;5(4):280-7. doi: 10.1046/j.1463-1318.2003.00497.x. PMID 12814403
- [Background] Rostaminia G, Abramowitch S, Chang C, Goldberg RP. The role of conventional pelvic floor reconstructive surgeries in obstructed defecation symptoms change: CARE and OPTIMAL trials sub-analysis of 2-year follow-up data. Int Urogynecol J. 2020 Jul;31(7):1325-1334. doi: 10.1007/s00192-019-04190-7. Epub 2019 Dec 24. PMID 31875258
- [Background] Bradley CS, Brown MB, Cundiff GW, Goode PS, Kenton KS, Nygaard IE, Whitehead WE, Wren PA, Weber AM; Pelvic Floor Disorders Network. Bowel symptoms in women planning surgery for pelvic organ prolapse. Am J Obstet Gynecol. 2006 Dec;195(6):1814-9. doi: 10.1016/j.ajog.2006.07.008. Epub 2006 Sep 25. PMID 16996465
- [Background] Bradley CS, Nygaard IE, Brown MB, Gutman RE, Kenton KS, Whitehead WE, Goode PS, Wren PA, Ghetti C, Weber AM; Pelvic Floor Disorders Network. Bowel symptoms in women 1 year after sacrocolpopexy. Am J Obstet Gynecol. 2007 Dec;197(6):642.e1-8. doi: 10.1016/j.ajog.2007.08.023. PMID 18060963
- [Background] Rostaminia G, Abramowitch S, Chang C, Goldberg RP. Descent and hypermobility of the rectum in women with obstructed defecation symptoms. Int Urogynecol J. 2020 Feb;31(2):337-349. doi: 10.1007/s00192-019-03934-9. Epub 2019 Apr 23. PMID 31016336
- [Background] Bordeianou L, Paquette I, Johnson E, Holubar SD, Gaertner W, Feingold DL, Steele SR. Clinical Practice Guidelines for the Treatment of Rectal Prolapse. Dis Colon Rectum. 2017 Nov;60(11):1121-1131. doi: 10.1097/DCR.0000000000000889. No abstract available. PMID 28991074
- [Background] Steele SR, Mellgren A. Constipation and obstructed defecation. Clin Colon Rectal Surg. 2007 May;20(2):110-7. doi: 10.1055/s-2007-977489. PMID 20011385
- [Background] Khaikin M, Wexner SD. Treatment strategies in obstructed defecation and fecal incontinence. World J Gastroenterol. 2006 May 28;12(20):3168-73. doi: 10.3748/wjg.v12.i20.3168. PMID 16718835
- [Background] VanderPas Lamb S, Massengill J, Sheridan MJ, Stern LE, von Pechmann W. Safety of combined abdominal sacral colpopexy and sigmoid resection with suture rectopexy: a retrospective cohort study. Female Pelvic Med Reconstr Surg. 2015 Jan-Feb;21(1):18-24. doi: 10.1097/SPV.0000000000000119. PMID 25185604
- [Background] Slawik S, Soulsby R, Carter H, Payne H, Dixon AR. Laparoscopic ventral rectopexy, posterior colporrhaphy and vaginal sacrocolpopexy for the treatment of recto-genital prolapse and mechanical outlet obstruction. Colorectal Dis. 2008 Feb;10(2):138-43. doi: 10.1111/j.1463-1318.2007.01259.x. Epub 2007 May 10. PMID 17498206
- [Background] Routzong MR, Abramowitch SD, Chang C, Goldberg RP, Rostaminia G. Obstructed Defecation Symptom Severity and Degree of Rectal Hypermobility and Folding Detected by Dynamic Ultrasound. Ultrasound Q. 2021 Sep 1;37(3):229-236. doi: 10.1097/RUQ.0000000000000565. PMID 34478420
- [Background] Rostaminia G, Abramowitch S, Chang C, Goldberg RP. Transvaginal sacrospinous ligament suture rectopexy for obstructed defecation symptoms: 1-year outcomes. Int Urogynecol J. 2021 Nov;32(11):3045-3052. doi: 10.1007/s00192-020-04611-y. Epub 2020 Nov 25. PMID 33237356
- [Background] Higgins PD, Johanson JF. Epidemiology of constipation in North America: a systematic review. Am J Gastroenterol. 2004 Apr;99(4):750-9. doi: 10.1111/j.1572-0241.2004.04114.x. PMID 15089911
- [Background] Blanchette G. The prevalence of pelvic floor disorders and their relationship to gender, age and mode of delivery. BJOG. 2003 Jan;110(1):88; author reply 88-9. doi: 10.1046/j.1471-0528.2003.01016_1.x. No abstract available. PMID 12504955
- [Background] Elshazly WG, El Nekady Ael A, Hassan H. Role of dynamic magnetic resonance imaging in management of obstructed defecation case series. Int J Surg. 2010;8(4):274-82. doi: 10.1016/j.ijsu.2010.02.008. Epub 2010 Feb 26. PMID 20219700
- [Background] Podzemny V, Pescatori LC, Pescatori M. Management of obstructed defecation. World J Gastroenterol. 2015 Jan 28;21(4):1053-60. doi: 10.3748/wjg.v21.i4.1053. PMID 25632177
- [Background] Kepenekci I, Keskinkilic B, Akinsu F, Cakir P, Elhan AH, Erkek AB, Kuzu MA. Prevalence of pelvic floor disorders in the female population and the impact of age, mode of delivery, and parity. Dis Colon Rectum. 2011 Jan;54(1):85-94. doi: 10.1007/DCR.0b013e3181fd2356. PMID 21160318

RESULTS

PARTICIPANT FLOW:
Groups:
- Unassigned: Due to early termination of the study, some enrolled participants remained as unassigned.
Period: Overall Study
Arm/Group | Laparoscopic Abdominal Ventral Rectopexy | Transvaginal Sacrospinous Rectopexy | Unassigned
Started | 5 | 6 | 4
Completed | 0 | 0 | 0
Not Completed | 5 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Unassigned: Due to the early termination of the study, some of the enrolled participants remained unassigned.
- Total: Total of all reporting groups
Arm/Group | Laparoscopic Abdominal Ventral Rectopexy | Transvaginal Sacrospinous Rectopexy | Unassigned | Total
Number analyzed (Participants) | 5 | 6 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (6.5) | 56.7 (8.9) | 59.5 (12.4) | 60.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 4 | 15
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 6 | 4 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 4 | 6 | 3 | 13
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Degree of Rectal Hypermobility Measured Via Ultrasound
Description: The degree of rectal hypermobility measured via ultrasound (i.e. compression ratio).
Time Frame: 24 months post-operatively
Population: Due to the early termination of the study, the 24-month post-operative primary outcome measurements could not be completed.
Arm/Group | Laparoscopic Abdominal Ventral Rectopexy | Transvaginal Sacrospinous Rectopexy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Postoperative Pain Measured by Pain Scale
Description: Participants will complete the pain scale. No pain will indicate the best outcome whereas the most intense pain imaginable will indicate the worst outcome.
Time Frame: 24 months post-operatively
Population: as for outcome 1
Arm/Group | Laparoscopic Abdominal Ventral Rectopexy | Transvaginal Sacrospinous Rectopexy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Postoperative Pain Measured by Pain Medication Use
Description: Participants will complete an assessment of pain medication use.
Time Frame: 24 months post-operatively
Population: as for outcome 1
Arm/Group | Laparoscopic Abdominal Ventral Rectopexy | Transvaginal Sacrospinous Rectopexy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Postoperative Functional Activity Level
Description: Participants will complete the Activity Assessment Scale which measures functional activity. The activity level will be measured on a scale of no difficulty, a little difficulty, some difficulty, a lot of difficulty, not able to do it, and did not do it for other reasons.
Time Frame: 24 months post-operatively
Population: as for outcome 1
Arm/Group | Laparoscopic Abdominal Ventral Rectopexy | Transvaginal Sacrospinous Rectopexy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Global Improvement in Bladder Function
Description: Participants will complete the Patient Global Impression of Improvement. The improvement will be measured on a scale of very much better, much better, a little better, no change, a little worse, much worse, and very much worse.
Time Frame: 24 months post-operatively
Population: as for outcome 1
Arm/Group | Laparoscopic Abdominal Ventral Rectopexy | Transvaginal Sacrospinous Rectopexy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Pelvic Floor Distress Inventory (PFDI) - POPDI
Description: As a part of the pelvic floor distress inventory (PFDI) questionnaire, participants will complete prolapse symptoms assessments using pelvic organ prolapse distress inventory (POPDI). The symptoms will be measured on a scale of 0, present, to 4, quite a bit. A higher score will indicate a higher symptom burden.
Time Frame: 24 months post-operatively
Population: as for outcome 1
Arm/Group | Laparoscopic Abdominal Ventral Rectopexy | Transvaginal Sacrospinous Rectopexy
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Pelvic Floor Distress Inventory (PFDI) - CRADI
Description: As a part of the pelvic floor distress inventory (PFDI) questionnaire, participants will complete colorectal symptoms assessments using colorectal anal distress inventory (CRADI). The symptoms will be measured on a scale of 0, present, to 4, quite a bit. A higher score will indicate a higher symptom burden.
Time Frame: 24 months post-operatively
Population: as for outcome 1
Arm/Group | Laparoscopic Abdominal Ventral Rectopexy | Transvaginal Sacrospinous Rectopexy
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Pelvic Floor Distress Inventory (PFDI) - UDI
Description: As a part of the pelvic floor distress inventory (PFDI) questionnaire, participants will complete urinary symptoms assessments using urinary distress inventory (UDI). The symptoms will be measured on a scale of 0, present, to 4, quite a bit. A higher score will indicate a higher symptom burden.
Time Frame: 24 months post-operatively
Population: as for outcome 1
Arm/Group | Laparoscopic Abdominal Ventral Rectopexy | Transvaginal Sacrospinous Rectopexy
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Quality of Life Measured by PFIQ
Description: Participants will complete pelvic floor impact questionnaire (PFIQ), a condition-specific health-related quality of life questionnaire. The measurement will be on a scale of 0, not at all, to 3, quite a bit. Higher scores indicate greater impact.
Time Frame: 24 months post-operatively
Population: as for outcome 1
Arm/Group | Laparoscopic Abdominal Ventral Rectopexy | Transvaginal Sacrospinous Rectopexy
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Quality of Life Measured by SF-36
Description: Participants will also complete short form health survey (SF-36), which measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). Higher scores indicate better health status.
Time Frame: 24 months post-operatively
Population: as for outcome 1
Arm/Group | Laparoscopic Abdominal Ventral Rectopexy | Transvaginal Sacrospinous Rectopexy
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Quality of Life Measured by EQ-5D
Description: Participants will complete EuroQol-5D (EQ-5D), an instrument that evaluates quality of life on five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The measurement will be on a scale of 1 to 5.
Time Frame: 24 months post-operatively
Population: as for outcome 1
Arm/Group | Laparoscopic Abdominal Ventral Rectopexy | Transvaginal Sacrospinous Rectopexy
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Pelvic Muscle Strength
Description: Participants will complete the Brink Scale, a digital assessment of pelvic floor muscle strength. It consists of 3 separate 4-point rating scales for pressure, vertical finger displacement, and duration.
Time Frame: 24 months post-operatively
Population: as for outcome 1
Arm/Group | Laparoscopic Abdominal Ventral Rectopexy | Transvaginal Sacrospinous Rectopexy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Laparoscopic Abdominal Ventral Rectopexy | Transvaginal Sacrospinous Rectopexy | Unassigned
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT05747027/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT05747027/ICF_001.pdf